CLINICAL TRIAL: NCT03503565
Title: The Effect of Intraoperative Neuromuscular Blockade on Postoperative Atelectasis in Patients Undergoing Thoracic Surgery With One Lung Ventilation: Moderate vs. Deep Block
Brief Title: Intraoperative Neuromuscular Blockade and Postoperative Atelectasis
Status: Completed | Type: Observational
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Hyungseok Seo, Clinical Associate Professor, Kyung Hee University Hospital at Gangdong
Other Study IDs: 2018-03-015
Record Dates: First submitted 2018-04-06; First posted 2018-04-20 (Actual); Results first posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Thoracic Surgery; One-lung Ventilation
Keywords: one-lung ventilation; thoracic surgery; atelectasis; postoperative pulmonary complication
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Moderate block group: maintaining moderate intraoperative neuromuscular blockade (TOF count 1 or 2) during surgery and reversal using sugammadex 2 mg/kg after surgery
  Interventions: Procedure: intraoperative neuromuscular blockade
- Deep block group: maintaining deep intraoperative neuromuscular blockade (PTC 1 or 2) during surgery and reversal using sugammadex 4 mg/kg after surgery
  Interventions: Procedure: intraoperative neuromuscular blockade

INTERVENTIONS:
Procedure: intraoperative neuromuscular blockade — The intensity of intraoperative neuromuscular blockade

SUMMARY:
During one-lung ventilation in thoracic surgery, the intensity of neuromuscular blockade may change the compliance and resistance of ventilated lung, thereby affecting postoperative atelectasis. The present study investigated the effect of the intensity of intraoperative neuromuscular blockade on the postoperative atelectasis using chest computerized tomography in patients receiving thoracic surgery requiring one-lung ventilation.

DETAILED DESCRIPTION:
Neuromuscular blocking agents can be used to secure a good surgical field, but it can also cause delayed extubation or postoperative pulmonary complications. Traditionally, rocuronium which is a commonly used non-depolarizing agent is usually reversed by cholinesterase inhibitors such as neostigmine or pyridostigmine. These drugs act by increasing the concentration of acetylcholine at the neuromuscular junction (a competing antagonist), not by direct antagonists. Consequently, there is a risk of pulmonary complications when cholinesterase inhibitor is not used appropriately. Use of sugammadex can reverse neuromuscular blockade (NMB) quickly, thereby being helpful for spontaneous deep breathing postoperatively. In a previous study, the moderate neuromuscular blockade was not guaranteed during surgery because intraoperative train-of-four (TOF) monitoring was not used and the outcome was focused on the correlation between reversal agent and the overall incidence of postoperative pulmonary complications. However, in the present study, TOF ratio or post-tetanic count (PTC) was repeatedly measured during surgery, thereby the intensity of intraoperative NMB being maintained. Moreover, lung compliance was repeatedly measured during surgery and the correlation between the intensity of intraoperative NMB and postoperative atelectasis which is evaluated by quantitative technique was also investigated.

Particularly in thoracic surgery, one lung ventilation is usually required for the surgical procedure. During one-lung ventilation, the compliance of ventilated lung is decreased and resistance can be increased, thereby the risk of atelectasis being increased. Furthermore, after thoracic surgery, although patients were encouraged to deep breathe, it is difficult to take a deep breath because of various factors. (i.e. pain, chest tube, long retracted time, postoperative interstitial edema, etc.) Therefore, postoperative atelectasis is much more important in patients undergoing thoracic surgery than other types of surgery.

For preventing postoperative atelectasis, the intraoperative intensity of neuromuscular blockade can be a crucial factor. Because deep neuromuscular blockade provides a good lung compliance during mechanical ventilation, peak inspiratory pressure can be decreased, thereby reducing the risk of ventilation-induced lung injury, particularly in one lung ventilation situation.However, there has been still lack of quantitative evidence that deep block is superior to moderate block in the thoracic surgery with one-lung ventilation

For assessment of postoperative atelectasis, plain chest radiography may be used. However, plain chest radiography can provide only a qualitative assessment of atelectasis. Computed tomography can assess the whole lung by its density (HU) and enables a quantitative assessment of postoperative atelectasis. Moreover, it can indicate the location of atelectasis more clearly than plain chest radiography, thus provide detailed information about postoperative lung state. To assess the effect of maintaining deep block and sugammadex reversal on the postoperative atelectasis, using chest CT can provide a much more quantitative and valuable information than conventional chest radiography.

ELIGIBILITY:
Inclusion Criteria:

1. Patients receiving scheduled unilateral lung lobectomy.
2. Patients age ≥19
3. Patients of American Society of Anesthesiologist Physical Status 1 or 2

Exclusion Criteria:

1. Patients receiving bilateral lung lobectomy
2. Patients BMI > 35.0 or < 18.5 kg/m2
3. Patients of contraindicated to epidural patients controlled analgesia
4. Patients with neuromuscular disease (i.e. myasthenia gravis)
5. Patients with major burn (more than 3rd degrees)
6. Patients with compromised cardiopulmonary function.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving open or thoracoscopic lobectomy, bi-lobectomy, or sleeve lobectomy.
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyungseok Seo, MD, PhD, Principal Investigator — Kyung Hee University Hospital at Gangdong
Locations (1):
- Kyung Hee University Gangdong Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho HC, Lee JH, Lee SC, Park SY, Rim JC, Choi SR. Use of sugammadex in lung cancer patients undergoing video-assisted thoracoscopic lobectomy. Korean J Anesthesiol. 2017 Aug;70(4):420-425. doi: 10.4097/kjae.2017.70.4.420. Epub 2017 Apr 21. PMID 28794837
- [Background] Grosse-Sundrup M, Henneman JP, Sandberg WS, Bateman BT, Uribe JV, Nguyen NT, Ehrenfeld JM, Martinez EA, Kurth T, Eikermann M. Intermediate acting non-depolarizing neuromuscular blocking agents and risk of postoperative respiratory complications: prospective propensity score matched cohort study. BMJ. 2012 Oct 15;345:e6329. doi: 10.1136/bmj.e6329. PMID 23077290
- [Background] Bulka CM, Terekhov MA, Martin BJ, Dmochowski RR, Hayes RM, Ehrenfeld JM. Nondepolarizing Neuromuscular Blocking Agents, Reversal, and Risk of Postoperative Pneumonia. Anesthesiology. 2016 Oct;125(4):647-55. doi: 10.1097/ALN.0000000000001279. PMID 27496656
- [Background] Casanova J, Pineiro P, De La Gala F, Olmedilla L, Cruz P, Duque P, Garutti I. [Deep versus moderate neuromuscular block during one-lung ventilation in lung resection surgery]. Rev Bras Anestesiol. 2017 May-Jun;67(3):288-293. doi: 10.1016/j.bjan.2017.02.005. Epub 2017 Feb 27. Portuguese. PMID 28256331
- [Background] Reinius H, Jonsson L, Gustafsson S, Sundbom M, Duvernoy O, Pelosi P, Hedenstierna G, Freden F. Prevention of atelectasis in morbidly obese patients during general anesthesia and paralysis: a computerized tomography study. Anesthesiology. 2009 Nov;111(5):979-87. doi: 10.1097/ALN.0b013e3181b87edb. PMID 19809292
- [Background] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A patient in Deep block group declined to participate in the study after enrollment.
Period: Overall Study
Arm/Group | Moderate Block Group | Deep Block Group
Started | 59 | 58
Completed | 59 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Block Group | Deep Block Group | Total
Number analyzed (Participants) | 59 | 58 | 117
Age, Customized [Median (Inter-Quartile Range); unit: years] | 64 [59 to 71] | 64 [58 to 73] | 64 [59 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 43 | 72
  Male | 30 | 15 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Preoperative abnormal chest radiography [Count of Participants; unit: Participants] — Population: Because the number of participants only counts the people who present abnormality on preoperative chest radiography
  Participants
    number analyzed (Participants) | 2 | 16 | 18
    Pleural effusion | 0 | 8 | 8
    Pneumothorax | 2 | 4 | 6
    Etc.(Pulmonary edema or infiltration, atelectasis, hemothrorax) | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Atelectasis Area on Chest CT
Description: Atelectasis on Chest CT The lung area was delineated manually. To calculate atelectasis, a region of interest was laid out that encircled the dense part of the lung, excluding large vessels. For further analysis, the lung was divided into four categories: areas with densities ranging from -1000 to -900 Hounsfield units (HU) were classified as over-aerated, from -900 to -500 HU as normally aerated, from -500 to -100 HU as poorly aerated, and from -100 to +100 HU as non-aerated (atelectasis). The proportion of non-aerated lung tissue (-100 to +100 HU) was calculated by dividing the area of the region of interest with the whole lungs.
Time Frame: 1 day after the end of surgery
Measure: Median (Inter-Quartile Range); unit: percentage of atelectasis volume
Arm/Group | Moderate Block Group | Deep Block Group
Number analyzed (Participants) | 58 | 56
percentage of atelectasis volume | 1.32 [0.47 to 3.20] | 1.41 [0.24 to 3.07]

2. Secondary Outcome: Number of Patients Defined as Acute Respiratory Distress Syndrome
Description: Acute respiratory distress syndrome can be defined as follows;
  Bilateral opacities not fully explained by effusions, lobar/lung collapse or nodules on chest radiograph or CT scan and Respiratory failure not fully explained by cardiac failure or fluid overload. Need objective assessment (e.g. echocardiography) to exclude hydrostatic edema if no risk factor present and Partial pressure of pulmonary arterial oxygen / Oxygen friction < 300 mmHg with positive end-expiratory pressure or continuous positive airway pressure of 5 cmH2O.
Time Frame: up to 7 days after the end of surgery
Reporting Status: Not Posted

3. Secondary Outcome: Number of Patients Defined as Pneumonia
Description: Pneumonia can be defined as follows;
  Two or more serial chest radiographs with at least one of the following (one radiograph is sufficient for patients with no underlying pulmonary or cardiac disease):
  1. new or progressive and persistent infiltrates
  2. consolidation
  3. cavitation; at least one of the following
  1) fever (>38.0 C) with no other recognized cause 2) White blood cell count < 4000/ml or >12,000/ml 3) for adults >70 yr, altered mental status with no other recognized cause; and at least two of the following
  1. new onset of purulent sputum or change in character of sputum, or increased respiratory secretions, or increased suctioning requirements
  2. new onset or worsening cough, or dyspnea, or tachypnea
  3. crackles or bronchial breath sounds
  4. worsening gas exchange (hypoxaemia, increased oxygen requirement, increased ventilator demand).
Time Frame: up to 7 days after the end of surgery
Reporting Status: Not Posted

4. Secondary Outcome: Number of Patients Showing Pleural Effusion
Description: Pleural effusion can be diagnosed on postoperative radiograph imaging.
Time Frame: 1 day after the end of surgery
Reporting Status: Not Posted

5. Secondary Outcome: Number of Patients Showing Postoperative Desaturation
Description: The number of patients showing desaturation (SpO2 <95%) in room air.
Time Frame: up to 1 day after surgery completed
Reporting Status: Not Posted

6. Secondary Outcome: Number of Patients Requiring Postoperative Re-intubation
Description: The number of patients requiring re-intubation due to postoperative respiratory difficulty.
Time Frame: up to 1 day after surgery completed
Reporting Status: Not Posted

7. Secondary Outcome: Intraoperative Lung Compliance (ml/cmH2O)
Description: Intraoperative lung compliance (ml/cmH2O) can be calculated with peak inspiratory pressure or plateau pressure, positive end-expiratory pressure and tidal volume.
Time Frame: every 1 hour from the time of the tracheal intubation to the end of the skin closure.
Reporting Status: Not Posted

8. Secondary Outcome: Patient Demographic Data
Description: Age in years, Gender, Weight in kilograms, Height in centimeters
Time Frame: on the day of admission
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 days
Description: All-Cause Mortality, Serious, or Other (non-serious) Adverse Events were monitored/assessed, but none observed.
Arm/Group | Moderate Block Group | Deep Block Group
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/58
Other Adverse Events (participants affected / at risk) | 0/59 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (1):
  • Study Protocol (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/65/NCT03503565/Prot_000.pdf